CLINICAL TRIAL: NCT01124435
Title: Phase II Study of the Combination Carboplatin Plus Celecoxib in Heavily Pre-treated Recurrent Ovarian Cancer Patients
Brief Title: Study of the Combination Carboplatin Plus Celecoxib in Heavily Pre-treated Recurrent Ovarian Cancer Patients
Acronym: carbo-cox2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Giovanni SCAMBIA-Department of Obstetrics and Gynecology-Catholic University of the Sacred Heart, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 935/03
Record Dates: First submitted 2010-05-14; First posted 2010-05-17 (Estimated); Last update posted 2010-06-04 (Estimated); Status verified 2008-12

CONDITIONS: Ovarian Neoplasms
Keywords: Carboplatin plus Celecoxib; Pre-treated Recurrent Ovarian Cancer Patients; The antitumor activity and potential adverse effects; tumor response rate; toxicity; progression free survival; duration of response; quality of life
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Carboplatin plus Celecoxib — celecoxib (200 mg tablets by mouth twice daily, day 1 to 28), associated to intravenous carboplatin (area under the curve (AUC) 5 over 30 to 60 minutes, every 28 days).

SUMMARY:
The aim of this study is to evaluate the antitumor activity and potential adverse effects of the combination celecoxib plus carboplatin in patients with recurrent, heavily pre-treated Ovarian Cancer (OC). The potential changes induced by the experimental combination on angiogenesis-related serum markers and quality of life measures will be also evaluated.The main objective is to evaluate the response rate. Secondary objectives are the following:toxicity;progression free survival;overall survival;duration of response;quality of life;modulation of angiogenesis-related molecules.

DETAILED DESCRIPTION:
This phase II prospective study will be conducted at the Gynecologic Oncology Units of the Catholic University of Rome and Campobasso, Italy. The study is non-sponsored, investigators initiated. The primary objective is to determine the tumor response rate by RECIST criteria. Secondary objectives included duration of response, progression-free survival (PFS), overall survival (OS), toxicity assessment, and QoL measures.Patients are required to take celecoxib (200 mg tablets by mouth twice daily, day 1 to 28), associated to intravenous carboplatin (area under the curve (AUC) 5 over 30 to 60 minutes, every 28 days). Patients who will develop carboplatin hypersensitivity reaction (HSR) will follow a desensitization protocol, or alternatively will switch to cisplatin. Erythropoietic stimulating agent and myeloid growth factors are not permitted for cycle 1 of study treatment, and their use will be chosen by the treating physician, according to hospital policy.Treatment will be discontinued when any of the following events occurs: radiographic or clinical evidence of cancer progression; deterioration of health or intolerable toxicity; patient refusal. Before starting treatment, patients will be evaluated by medical history, physical examination, cell blood count (CBC), chemistry panel, Ca125, and either computed tomography or magnetic resonance imaging scan. The primary endpoint is to determine the overall response (OR) rate. Secondary endpoints include the assessment of duration of response, PFS, OS, toxicity events and QoL scores. When treatment will be discontinued, patients will receive a follow-up visit every 3 months

ELIGIBILITY:
Inclusion Criteria:

* Recurrent epithelial ovarian or fallopian tube or peritoneal serous carcinomas with measurable disease as assessed by Response Evaluation Criteria in Solid Tumors criteria
* Patients will require to have received a platinum-containing regimen as primary treatment and at least one line of chemotherapy for recurrent disease
* An interval time from the last platinum-based chemotherapy after 6months
* 18 years of years
* Eastern Cooperative Oncology Group performance status of 0 to 2
* Adequate bone marrow
* Adequate renal and hepatic functions
* Written informed consent to the study protocol

Exclusion Criteria:

* Hypersensitivity to celecoxib or aspirin or other nonsteroidal anti-inflammatory drugs or sulfonamides
* Significant comorbidities including any active coronary artery disease requiring management or symptomatic congestive heart failure or bleeding diathesis or uncontrolled severe hypertension or active gastrointestinal ulcer within 12 months or chronic inflammatory bowel diseases or deep venous or arterial thrombosis within 12 months or history of pulmonary embolism
* Concomitant use of possible interactive drugs
* Surgery and chemotherapy or radiotherapy within 1 month
* Actual or potential childbearing
* Breast-feeding
* Prior cancer treatment with a COX2 inhibitor
* Any psychological and/or sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-10; Primary Completion 2007-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of the Combination Carboplatin plus Celecoxib in Heavily Pre-treated Recurrent Ovarian Cancer Patients | 48 months
  The tumor response rate by Response Evaluation Criteria in Solid Tumors (RECIST) criteria and duration of response, progression-free survival (PFS), overall survival (OS), toxicity assessment, and quality of life (QoL) measures with carboplatin-celcoxib in heavly pretreated recurrent ovarian cancer patients.

SECONDARY OUTCOMES:
The modulation of angiogenesis-related molecules with the combination celecoxib plus carboplatin in patients with recurrent, heavily pre-treated OC | 12 months
  Serum levels of vascular endothelial growth factor (VEGF) and endostatin evaluated in a preliminary series of 11 patients at baseline and after 1 month of carboplatin-celecoxib

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni sCAMBIA, PhD, Principal Investigator — Department of Obstetrics and Gynecology,
Locations (1):
- Department of Obstetrics and Gynecology,Catholic University, Rome, Italy, Rome, Italy, Italy

REFERENCES:
- [Result] Ferrandina G, Lauriola L, Zannoni GF, Fagotti A, Fanfani F, Legge F, Maggiano N, Gessi M, Mancuso S, Ranelletti FO, Scambia G. Increased cyclooxygenase-2 (COX-2) expression is associated with chemotherapy resistance and outcome in ovarian cancer patients. Ann Oncol. 2002 Aug;13(8):1205-11. doi: 10.1093/annonc/mdf207. PMID 12181243
- [Derived] Legge F, Paglia A, D'Asta M, Fuoco G, Scambia G, Ferrandina G. Phase II study of the combination carboplatin plus celecoxib in heavily pre-treated recurrent ovarian cancer patients. BMC Cancer. 2011 May 31;11:214. doi: 10.1186/1471-2407-11-214. PMID 21627839